CLINICAL TRIAL: NCT00757289
Title: Use of Platelet-rich-plasma to Treat Tennis Elbow, A Blinded and Randomized Single Center Study
Brief Title: Platelet-rich-plasma Treating Tennis Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMET NL 03
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: Tennis Elbow
MeSH Terms: conditions — Pain; Tennis Elbow | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PRP injection
  Interventions: Biological: PRP Injection
- 2 (Active Comparator): Corticosteroid Injection
  Interventions: Biological: Corticosteroid Injection

INTERVENTIONS:
Biological: PRP Injection — PRP Injection
  Arms: 1
Biological: Corticosteroid Injection — Corticosteroid Injection
  Arms: 2

SUMMARY:
The study is to compare the efficacy of autologous platelet concentrate injections to corticosteroid injection in patients suffering from tennis elbow with respect to pain and function.

DETAILED DESCRIPTION:
Patients with chronic plantar fasciitis will be allocated randomly to have a steroid injection or an autologous platelet concentrate injections. Data will be collected before the procedure, 4, 8, 12, 26 weeks and 1 year after the procedure. The main outcome measures of this study are pain and function measured with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic epicondylitis lateralis who do not react to conservative treatment and therefore are send to the orthopedic surgeon

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Score - Pain | 4months,12 months,24months & 52 months

SECONDARY OUTCOMES:
DASH | 4months,12months,24months & 52 months
Complications | Anytime

CONTACTS AND LOCATIONS:
Overall Officials: Taco Gosens, MD, Principal Investigator — Elisabeth ziekenhuis
Locations (1):
- Elisabeth ziekenhuis, Tilburg, Netherlands

IPD SHARING:
Plan to Share IPD: No